CLINICAL TRIAL: NCT03207165
Title: Comparison of Milrinone Versus Dobutamine in a Heterogeneous Population of Critically Ill Patients
Brief Title: Milrinone Versus Dobutamine in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160975-01H
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Low Cardiac Output Syndrome; Cardiogenic Shock; Acute Coronary Syndrome; Pulmonary Edema
Keywords: Cardiogenic shock; Inotropes; Low cardiac output syndrome
MeSH Terms: conditions — Cardiac Output, Low; Shock, Cardiogenic; Acute Coronary Syndrome; Pulmonary Edema | interventions — Milrinone; N(1)-methyl-2-lysergic acid diethylamide; Dobutamine

STUDY DESIGN:
Intervention Model Description: Consecutive patients admitted to the Coronary Care Unit (CCU) at the Ottawa Heart Institute from start of study (tentatively set for August 2017 with anticipated end date of June 2020) and identified by the treating medical team as requiring initiation of inotrope therapy will be screened and randomized based on the healthcare team's clinical assessment of predominantly LV or RV systolic dysfunction (biventricular dysfunction will be assigned to predominantly LV dysfunction). All decisions to initiate inotrope therapy will be made by the primary care team with no involvement from the research team.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study participants, treating medical team and research team will be blinded to randomization; the pharmacy staff, CCU nurses and allied healthcare team members will not be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left ventricular [LV] +/- Biventricular dysfunction (Active Comparator): Assessment of left ventricular [LV] or biventricular dysfunction will be based on clinical assessment, available imaging (echocardiogram, left ventriculogram, MUGA/RNA scan, cardiac MRI, etc.) and known past medical history (if available and contributory). Patients identified as having biventricular dysfunction will be randomized within the LV dysfunction arm of the trial. Patients in this arm will be randomized in a 1:1 fashion to Milrinone or Dobutamine.
  Interventions: Drug: Milrinone; Drug: Dobutamine
- Right ventricular [RV] dysfunction (Active Comparator): Assessment of right ventricular [RV] dysfunction will be based on clinical assessment, available imaging (echocardiogram, left ventriculogram, MUGA/RNA scan, cardiac MRI, etc.) and known past medical history (if available and contributory). Patients in this arm will be randomized in a 1:1 fashion to Milrinone or Dobutamine.
  Interventions: Drug: Milrinone; Drug: Dobutamine

INTERVENTIONS:
Drug: Milrinone — Patients will be initiated on Milrinone at 0.125 mcg/kg/min [stage 1] and will be titrated according to a blinded protocol from stages 2 to 5 [0.250, 0.375, 0.5 and >0.5 ug/kg/min]. All orders to initiate and titrate the dose of the allocated inotrope will be written in the chart as follows: 'Study inotrope dose to be [increased/decreased/maintained] at stage [1-5]' so as to ensure that treating physicians remain blinded to the allocated drug.
  Other Names: Mil; Phosphodiesterase-3 inhibitors [PDE3] Inhibitor
Drug: Dobutamine — Patients will be initiated on Dobutamine at 2.5 mcg/kg/min [stage 1] and will be titrated according to a blinded protocol from stages 2 to 5 [5.0, 7.5, 10 and >10 ug/kg/min]. All orders to initiate and titrate the dose of the allocated inotrope will be written in the chart as follows: 'Study inotrope dose to be [increased/decreased/maintained] at stage [1-5]' so as to ensure that treating physicians remain blinded to the allocated drug.
  Other Names: Dob; Beta 1/2 Agonist

SUMMARY:
The investigators are interested in determining if there is a meaningful difference between two of the most commonly used medications used to improve the pumping function of the heart among critically ill patients admitted to the Coronary Care Unit (CCU) at the University of Ottawa Heart Institute (UOHI). To do this, the investigators will randomly assign patients who are felt to require use of these medications by their treating physicians to one of the two most commonly used agents in Canada: Milrinone or Dobutamine. Each patient will be closely monitored by their healthcare team, and their medication will be adjusted based on each patient's clinical status. Information from blood work (e.g. kidney and liver function, complete blood counts, and other markers of how effectively blood is circulating in the body), assessment of end-organ function (e.g. urine output, mentation), abnormal heart rhythms noted on monitoring and results of imaging studies (e.g. angiogram, echocardiograms.) will be collected for analysis. All patients will be followed for the duration of their hospital stay at UOHI.

DETAILED DESCRIPTION:
The use of various inotropes in the care of critically ill cardiac patients has become increasingly widespread: while predominantly used in decompensated heart failure, they have also been used in cardiogenic shock complicating acute coronary syndrome (ACS) and septic shock. Purported mechanisms of efficacy include improved cardiac output, improved end-organ perfusion, and vasodilation of both pulmonary and systemic circulations. Two of the most commonly used agents are Milrinone, a phosphodiesterase 3 inhibitor, and Dobutamine, a synthetic catecholamine with affinity for both beta-1 and 2 receptors. Both the American College of Cardiology (ACC) and the European Society of Cardiology (ESC) support inotropes for acute and chronic heart failure management with low cardiac output states. Furthermore, the ACC recommends consideration of inotropic therapy within the STEMI guidelines when ACS is complicated by cardiogenic shock, heart failure or for hemodynamic support in isolated right ventricle infarctions. Beyond primarily cardiac etiologies, inotropes have been identified as first-line additive therapy for cardiac augmentation to Norepinephrine in patients with septic shock complicated by myocardial dysfunction. Despite the lack of convincing data supporting a morbidity or mortality benefit with the use of inotropes in severe, decompensated heart failure, cardiogenic or septic shock, or in ACS, inotropic therapy is still widely used across various critical care settings. Furthermore, to date, there has been no head to head comparison of the two more commonly used positive inotropes: Dobutamine and Milrinone. Selection of one inotrope over another is often guided by physician and center preference, and consideration of and purported avoidance of possible adverse effects. In this pilot study, the investigators aim to describe that characteristics of patients receiving inotropic support in the CCU setting and identify possible differences in morbidity and mortality between Dobutamine and Milrinone among a heterogeneous population of patients admitted to the CCU at UOHI, which may help to inform a larger clinical trial in the future.

The purpose of this pilot study is to: (a) describe the characteristics of patients receiving inotropic support in the coronary care unit (CCU) setting (hemodynamics prior to inotrope initiation, etiology of cardiogenic shock state, use of PA catheter and values if deemed necessary by medical team) and (b) identify possible differences in morbidity [atrial and ventricular arrhythmias, hepatic and renal function, markers of end-organ perfusion (lactate, urine output, mentation status), use of vasopressors, sustained hypotension of systolic blood pressure less than or equal to 90 mmHg for greater than 30 minutes, need for mechanical support, cardiac transplant, total length of CCU stay, length of CCU stay greater than 14 days] and mortality between patients in cardiogenic shock treated with Dobutamine versus Milrinone.

ELIGIBILITY:
Inclusion Criteria:

* Have one or more of the following:
* Low cardiac output state, evidenced by sustained hypotension (systolic blood pressure <90 mmHg) and end organ dysfunction (altered level of consciousness, elevated lactate, renal or hepatic dysfunction)
* Clinical evidence of systemic and/or pulmonary congestion despite use of vasodilators and/or diuretics
* ACS complicated by cardiogenic shock (defined as persistent hypotension with systolic blood pressure <90 mmHg with severe reduction in cardiac index [<1.8 L/min/m2 without support or <2.2 L/min/m2 with support], left ventricular end-diastolic pressure >18 mmHg)
* Augmentation of cardiac output when patient already on maximal vasopressor therapy
* Or medical team's decision that patient needs inotropic therapy

Exclusion Criteria:

* Unwillingness or inability to provide informed consent by the patient or substitute decision maker for healthcare decisions
* Female participants who are currently pregnant
* Patients presenting with an out-of-hospital cardiac arrest (OOHCA)
* Healthcare team preference for use of specific inotrope (Milrinone or Dobutamine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Composite Primary End Point | Through duration of hospitalization, up to 12 weeks following admission
  Composite of all-cause in-hospital death, non-fatal MI, TIA or CVA diagnosed by a Neurologist, renal failure requiring renal replacement therapy, need for cardiac transplant or new mechanical support, any atrial or ventricular arrhythmia leading to cardiac arrest and resuscitation.
All-cause in-hospital death | Through duration of hospitalization, up to 12 weeks following admission
  All-cause in-hospital death
Non-fatal myocardial infarction [MI] | Through duration of hospitalization, up to 12 weeks following admission
  As defined by Thygesen et al., 2012 (Circulation)
Transient ischemic attack [TIA] or cerebrovascular accident [CVA] | Through duration of hospitalization, up to 12 weeks following admission
  Transient ischemic attack or cerebrovascular accident as diagnosed by a Neurologist either clinically and/or radiographically
Stay in CCU greater than or equal to 7 days | Through duration of hospitalization, up to 12 weeks following admission
  Stay in CCU greater than or equal to 7 days
Acute kidney injury requiring renal replacement therapy | Through duration of hospitalization, up to 12 weeks following admission
  Acute kidney injury requiring renal replacement therapy (intermittent hemodialysis or continuous renal replacement therapy)
Need for advanced mechanical support [specifically, intra-aortic balloon pump, Impella, ventricular assist device or extra-corporeal membrane oxygenation] or cardiac transplant | Through duration of hospitalization, up to 12 weeks following admission
  Need for new mechanical support or cardiac transplant

SECONDARY OUTCOMES:
Time on inotropes | Through duration of hospitalization, up to 12 weeks following admission
  Total time on inotropes (in hours)
Non-invasive or invasive mechanical ventilation | Through duration of hospitalization, up to 12 weeks following admission
  Total number of days requiring non-invasive or invasive mechanical ventilation
Change in cardiac index ([CI] | Through duration of hospitalization, up to 12 weeks following admission
  Change in cardiac index measured with PA catheter
Change in pulmonary capillary wedge pressure [PCWP] | Through duration of hospitalization, up to 12 weeks following admission
  Change in pulmonary capillary wedge pressure measured with PA catheter
Change in pulmonary vascular resistance [PVR] | Through duration of hospitalization, up to 12 weeks following admission
  Change in pulmonary vascular resistance measured with PA catheter
Change in systemic vascular resistance [SVR] | Through duration of hospitalization, up to 12 weeks following admission
  Change in systemic vascular resistance measured with PA catheter
Presence of acute kidney injury | Through duration of hospitalization, up to 12 weeks following admission
  Presence of acute kidney injury (defined by KDIGO as creatinine increased by 26.5 umol/L, 1.5 times baseline within prior 7 days, or urine volume <0.5 mL/kg/hour for greater than or equal to 6 hours
Serum lactate | Through duration of hospitalization, up to 12 weeks following admission
  Normalization of serum lactate
Arrhythmia requiring medical team intervention | Through duration of hospitalization, up to 12 weeks following admission
  Arrhythmia requiring medical team intervention, either through electrical or chemical cardioversion or any intravenous anti-arrhythmia medication administration

OTHER OUTCOMES:
Sustained hypotension of systolic BP | Through duration of hospitalization in CCU, up to 12 weeks following admission
  Sustained systolic blood pressure hypotension of less than or equal to 90 mmHg for greater than or equal to 30 minutes (or requiring medical intervention)
Atrial arrhythmias requiring medical intervention | Through duration of hospitalization in CCU, up to 12 weeks following admission
  Atrial flutter, fibrillation or tachycardia requiring medical intervention
Need for intravenous or oral anti-arrhythmic therapy | Through duration of hospitalization in CCU, up to 12 weeks following admission
  Initiation of intravenous or oral anti-arrhythmic therapy
Ventricular arrhythmias | Through duration of hospitalization in CCU, up to 12 weeks following admission
  Ventricular arrhythmias (monomorphic or polymorphic ventricular tachycardia [VT] greater than 30 seconds or hemodynamically unstable ventricular arrhythmia requiring intervention, or VF)
Need for up-titration or addition of new vasopressor therapy | Through duration of hospitalization in CCU, up to 12 weeks following admission
  Need for up-titration or addition of new vasopressor therapy

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Hibbert, MD, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abraham WT, Adams KF, Fonarow GC, Costanzo MR, Berkowitz RL, LeJemtel TH, Cheng ML, Wynne J; ADHERE Scientific Advisory Committee and Investigators; ADHERE Study Group. In-hospital mortality in patients with acute decompensated heart failure requiring intravenous vasoactive medications: an analysis from the Acute Decompensated Heart Failure National Registry (ADHERE). J Am Coll Cardiol. 2005 Jul 5;46(1):57-64. doi: 10.1016/j.jacc.2005.03.051. PMID 15992636
- [Background] Aranda JM Jr, Schofield RS, Pauly DF, Cleeton TS, Walker TC, Monroe VS Jr, Leach D, Lopez LM, Hill JA. Comparison of dobutamine versus milrinone therapy in hospitalized patients awaiting cardiac transplantation: a prospective, randomized trial. Am Heart J. 2003 Feb;145(2):324-9. doi: 10.1067/mhj.2003.50. PMID 12595851
- [Background] Karlsberg RP, DeWood MA, DeMaria AN, Berk MR, Lasher KP. Comparative efficacy of short-term intravenous infusions of milrinone and dobutamine in acute congestive heart failure following acute myocardial infarction. Milrinone-Dobutamine Study Group. Clin Cardiol. 1996 Jan;19(1):21-30. doi: 10.1002/clc.4960190106. PMID 8903534
- [Background] King JB, Shah RU, Sainski-Nguyen A, Biskupiak J, Munger MA, Bress AP. Effect of Inpatient Dobutamine versus Milrinone on Out-of-Hospital Mortality in Patients with Acute Decompensated Heart Failure. Pharmacotherapy. 2017 Jun;37(6):662-672. doi: 10.1002/phar.1939. PMID 28475215
- [Background] Yamani MH, Haji SA, Starling RC, Kelly L, Albert N, Knack DL, Young JB. Comparison of dobutamine-based and milrinone-based therapy for advanced decompensated congestive heart failure: Hemodynamic efficacy, clinical outcome, and economic impact. Am Heart J. 2001 Dec;142(6):998-1002. doi: 10.1067/mhj.2001.119610. PMID 11717603
- [Derived] Marbach JA, Di Santo P, Kapur NK, Thayer KL, Simard T, Jung RG, Parlow S, Abdel-Razek O, Fernando SM, Labinaz M, Froeschl M, Mathew R, Hibbert B. Lactate Clearance as a Surrogate for Mortality in Cardiogenic Shock: Insights From the DOREMI Trial. J Am Heart Assoc. 2022 Mar 15;11(6):e023322. doi: 10.1161/JAHA.121.023322. Epub 2022 Mar 9. PMID 35261289
- [Derived] Jung RG, Di Santo P, Mathew R, Abdel-Razek O, Parlow S, Simard T, Marbach JA, Gillmore T, Mao B, Bernick J, Theriault-Lauzier P, Fu A, Lau L, Motazedian P, Russo JJ, Labinaz M, Hibbert B. Implications of Myocardial Infarction on Management and Outcome in Cardiogenic Shock. J Am Heart Assoc. 2021 Nov 2;10(21):e021570. doi: 10.1161/JAHA.121.021570. Epub 2021 Oct 29. PMID 34713704
- [Derived] Di Santo P, Mathew R, Jung RG, Simard T, Skanes S, Mao B, Ramirez FD, Marbach JA, Abdel-Razek O, Motazedian P, Parlow S, Boczar KE, D'Egidio G, Hawken S, Bernick J, Wells GA, Dick A, So DY, Glover C, Russo JJ, McGuinty C, Hibbert B; CAPITAL DOREMI investigators. Impact of baseline beta-blocker use on inotrope response and clinical outcomes in cardiogenic shock: a subgroup analysis of the DOREMI trial. Crit Care. 2021 Aug 10;25(1):289. doi: 10.1186/s13054-021-03706-2. PMID 34376218
- [Derived] Mathew R, Di Santo P, Jung RG, Marbach JA, Hutson J, Simard T, Ramirez FD, Harnett DT, Merdad A, Almufleh A, Weng W, Abdel-Razek O, Fernando SM, Kyeremanteng K, Bernick J, Wells GA, Chan V, Froeschl M, Labinaz M, Le May MR, Russo JJ, Hibbert B. Milrinone as Compared with Dobutamine in the Treatment of Cardiogenic Shock. N Engl J Med. 2021 Aug 5;385(6):516-525. doi: 10.1056/NEJMoa2026845. PMID 34347952